CLINICAL TRIAL: NCT05647889
Title: Investigation of the Effect of Jet Lidocaine and Ice Application on Reduction of Pain and Anxiety Related to Peripheral Venous Catheterisation in Adult Patients: A Randomised Controlled Trial
Brief Title: Pain and Anxiety in Peripheral Venous Catheterization, Jet Lidocaine, Ice Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Esra Aydın, Lecturer, Ataturk University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: ATATURKUNIVERSITYESRAAYDIN0029
Record Dates: First submitted 2022-10-20; First posted 2022-12-13 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Peripheral Venous Catheterization
Keywords: Pain; Anxiety; Ice application; Jet Lidocaine; Nursing; Peripheral venous catheterization
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Ice

STUDY DESIGN:
Intervention Model Description: In the study, 80 individuals, including 2 experimental and 1 control group, were included in the study.
Who Masked: Care Provider
Masking Description: To control the research in terms of bias; During the data collection phase, help will be taken from the clinical nurse who takes care of the patient. The nurse, who does not know which intervention is applied, will be asked to evaluate the patient's pain and anxiety. In this respect, the research will be considered single-blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Jet lidocaine group (Experimental): Jet lidocaine will be applied before PVC and PVC will be performed 3 minutes later.
  Interventions: Drug: Jet lidocaine
- Ice group (Experimental): Ice will be applied for 1 minute before PVC, and then PVC will be performed.
  Interventions: Combination Product: Ice
- Control group (Active Comparator): Standard PVC procedure will be applied
  Interventions: Other: Standard PVC procedure

INTERVENTIONS:
Drug: Jet lidocaine — Jet lidocaine will be applied before PVC and PVC will be performed 3 minutes later.
  Other Names: Intervention group-I
  Arms: Jet lidocaine group
Combination Product: Ice — Ice will be applied for 1 minute before PVC, and then PVC will be performed.
  Other Names: Intervention group-II
  Arms: Ice group
Other: Standard PVC procedure — Standard PVC procedure will be applied
  Other Names: standard application group
  Arms: Control group

SUMMARY:
Investigation of the Effect of Jet Lidocaine and Ice Application on Pain and Anxiety in Peripheral Venous Catheterization (PVC). The research will be carried out experimentally with a single group post-test method. The universe of the research; Between June-December 2022, all patients who need peripheral venous catheterization (PVK) for the treatment plan will be formed in the internal clinics of Gümüşhane State Hospital. The sample of the study will consist of 80 patients from the defined population who meet the inclusion criteria. Power analysis was used to determine the number of samples in the study. First of all, patients who are hospitalized in the internal clinics of Gümüşhane State Hospital and who meet the inclusion criteria will be determined. Written and verbal consent will be obtained for their participation by giving information about the research. PVK application will be applied to all patients by the same investigator. Each patient will create their own control group in order to control individual differences in pain and anxiety. In the study consisting of two intervention and a control group; The same patients will be included in the intervention groups and the control group. Randomization will be done to determine the order of intervention to be applied to the patients. The interventions for each patient will be numbered by the researcher and the order of procedure will be determined by drawing lots. After the cephalic vein for the first attempt is randomly determined, the other extremity vein will be used while performing consecutive PVC applications. To control the research in terms of bias; During the data collection phase, help will be taken from the clinical nurse who takes care of the patient. The nurse, who does not know which intervention is applied, will be asked to evaluate the patient's pain and anxiety. In this respect, the research will be considered single-blind.

DETAILED DESCRIPTION:
This study was planned as a randomized controlled, single-blind experiment. The research will be carried out in the internal clinics of Gümüşhane State Hospital. Internal clinics were preferred because patients hospitalized in surgical clinics experienced intense pain and anxiety due to surgical operations. The universe of the research; All patients who are hospitalized in the relevant clinics within the specified time period and who need to apply PVC for the treatment plan will be formed.

The sample of the research; It will consist of 80 patients who are hospitalized in internal clinics, who need PVC for diagnosis or treatment, and who meet the research criteria. Power analysis was used to determine the number of samples in the study.The data of the research; Patient Information Form will be collected using the Visual Analog Scale for Pain (VAS-P), Visual Analog Scale for Anxiety (VAS-A), Wong-Baker Faces Pain Rating Scale. Nursing Intervention: The research will be conducted experimentally with a single group post-test method. First of all, patients who meet the criteria for inclusion in the study will be determined, and written and verbal consent will be obtained for their participation by giving information about the research. PVC application will be applied to all patients by the same investigator. Each patient will create their own control group in order to control individual differences in pain and anxiety. In the study consisting of two intervention and a control group; The same patients will be included in the intervention groups and the control group. Randomization will be done to determine the order of intervention to be applied to the patients. Interventions will be numbered for each patient and the order of procedure will be determined by drawing lots. After the cephalic vein for the first attempt is randomly determined, the other extremity vein will be used while performing consecutive PVC applications. To control the research in terms of bias; During the data collection phase, help will be taken from the clinical nurse who takes care of the patient. The nurse, who does not know which intervention is applied, will be asked to evaluate the patient's pain and anxiety. In this respect, the research will be considered single-blind.

Intervention group-I (Jet lidocaine will be applied before PVC and PVC will be performed 3 minutes later) Intervention group-II (Ice application will be made for 1 minute before PVC and then PVC will be performed) It will be named as the control group (Standard PVC procedure will be applied)

Process steps

Control group PVC Application Steps

1. Hands will be washed.
2. The treatment tray will be prepared.
3. The correct patient will be determined, the procedure will be explained to the patient and permission will be obtained.
4. A "Patient Identification Form" will be applied to the individual before PVC.
5. The individual will be given a fowler, semi fowler or supine position.
6. The area where PVC will be applied will be checked for phlebitis, thrombophlebitis, ecchymosis, hematoma and signs of local infection.
7. The vein to be administered will be evaluated by observing and palpating in terms of intervention.
8. By wearing gloves, the side grip sections of the peripheral venous catheter (22 G) will be brought to the horizontal position.
9. A tourniquet will be attached 10-15 cm above the area where the catheter will be entered.
10. The catheter will be held between the thumb and forefinger with the tapered side of the needle facing up.
11. The individual will be asked to turn their head in the opposite direction to the side where the peripheral venous catheter will be inserted.
12. Cleaning of the area will be done with a cotton pad with antiseptic in a single movement in the direction of arterial blood circulation and it will be waited for about 5 seconds for the area to dry.
13. The catheter will be held at an angle of 30-45° to the skin, approximately 1 cm below the area where the vein is to be entered, and the vein will be accessed.
14. As soon as the needle enters the vein, it will be slowly advanced into the vein, reducing the angle to approximately 15°.
15. It will be checked whether there is blood coming to the blood stopper valve and if there is blood, the catheter will continue to be advanced in the vein.
16. At this stage, the needle of the catheter will be withdrawn with the passive hand, while the plastic part will be advanced into the vein with the active hand simultaneously.
17. The level of pain related to the PVC application during the insertion of the catheter will be evaluated by the clinical nurse with the Wong-Baker Faces Pain Rating Scale.
18. Without moving the catheter in the vein, the tourniquet will be loosened with the inactive hand, fixed temporarily with a small patch, the needle of the catheter will be removed and the cap of the catheter will be closed.
19. Permanent fixation of the catheter will be performed.
20. Contaminated materials will be removed from the environment.
21. Within 1 minute after catheter placement, patients' pain and anxiety levels related to PVC application will be evaluated with VAS-A and VAS-P.

Intervention group-I PVC Application Steps

1. Implementation steps 1-7 of the Control Group will be done.
2. A tourniquet will be tied 10-15 cm above the area where the catheter will be inserted by wearing gloves.
3. After the area to be intervened is determined, the tourniquet will be dissolved, the area will be cleaned with a cotton pad with antiseptic from top to bottom in a single movement, and the area will be waited for 5 seconds to dry.
4. The dermis layer on the vein determined for intervention will be pulled to the side with the help of the passive hand (without any venous intervention), and the head of the lidocaine-loaded jet device will be firmly placed on the cit at an angle of 90°.
5. Since 0.3 ml of lidocaine solution or 3 mg of total dose will not pose a problem in terms of drug toxicity; 0.3 ml 1% lidocaine will be applied with a Jet device and waited for 5 seconds.
6. After waiting for 5 seconds, the Jet device will be lifted and the skin will be released.
7. Catheter intervention will be performed after 3 min to achieve optimal anesthetic conditions.
8. The lateral grips of the peripheral venous catheter (22 G) will be placed in the horizontal position.
9. The process will be completed by performing the steps between 9-11 and 13-21 of the Control Group.

Initiative Group-II PVC Application Steps

1. Implementation steps of the Control Group 1-7 will be done.
2. In order to create an anesthetic effect; Ice will be applied for 1 minute to the designated area to enter before PVC.
3. The process will be completed by performing the 8-21 application steps of the Control Group.Variables of the Study Dependent variables were: Visual Analog Scale Score for Anxiety (VAS-A), Visual Analog Scale Score for Pain (VAS-P), and Wong-Baker Faces Pain Rating Scale Score.

Independent variables:

0.3 ml Jet lidocaine application before peripheral venous catheterization

1 minute ice application before peripheral venous catheterization

Control variables:

Peripheral venous catheterization site (Cephalic vein), Catheter diameter and length (22 G)

Evaluation of data: The data will be evaluated in the SPSS (Statistical Package for Social Sciences for Windows, Version 22.0) package program. In the evaluation of the data, the statistical significance value will be accepted as 0.05, the Type 1 error will be kept at 5% and the evaluation will be made with a 95% confidence interval

ELIGIBILITY:
Inclusion Criteria:

1. Able to speak and understand Turkish,
2. Those between the ages of 18-50,
3. Demanding peripheral venous catheter insertion,
4. Having lidocaine request before PVC,
5. Having no problems with vision and hearing,
6. No history of secondary acute pain other than peripheral venous catheter,
7. Having no physical barrier to insertion of a catheter from the cephalic veins,
8. Not allergic to lidocaine and cold,
9. No signs of phlebitis, scar tissue, dermatitis, incision and infection in the area to be operated,
10. No history of peripheral nerve disease, peripheral neuropathy, paresis, plegia or hemiplegia that may affect the sensation of pain,
11. Individuals without coagulation disorder, liver failure, kidney and cardiovascular failure will be included in the study.

Exclusion Criteria:

1. Cannot speak or understand Turkish,
2. Those who are outside the age range of 18-50,
3. No request for peripheral venous catheter insertion,
4. No lidocaine request before PVC,
5. Having any problems with vision and hearing,
6. Having a history of any secondary acute pain other than peripheral venous catheter,
7. Having a physical obstacle to insertion of a catheter from the cephalic veins,
8. Those who are allergic to lidocaine and cold,
9. With phlebitis, scar tissue, dermatitis, incision and infection findings in the area to be operated,
10. Having a history of peripheral nerve disease, peripheral neuropathy, paresis, plegia or hemiplegia that may affect the sensation of pain,
11. Patients with coagulation disorder, liver failure, kidney and cardiovascular failure

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale for Pain (VAS-P) | Within 1 minute after PVC application
  It is a scale used to evaluate the severity of pain. It is a 100 mm ruler with painlessness at one end and the most severe pain at the other. "0" denotes painlessness, and "100" denotes the most severe pain.A low score from the scale indicates that the application is beneficial.

SECONDARY OUTCOMES:
Visual Analogue Scale for Anxiety (VAS-A) | Within 1 minute after PVC application
  VAS-A; It consists of a continuous horizontal line 0-100 mm long. "0" represents I am not nervous at all, while "100" represents I am extremely nervous. Participants indicate their level of anxiety by specifying a position between the two extremes.A low score from the scale indicates that the application is beneficial.

OTHER OUTCOMES:
Wong-Baker Faces Pain Rating Scale | While performing the PVC application
  The revised version of the scale is widely used in the assessment of pain severity in the adult and pediatric population. The scale includes visual representations of six facial expressions that increasingly represent pain intensity. Pain score is given according to the numerical values given to the faces in the scale. The lowest score is "0" and the highest score is "10". As the score obtained from the scale increases, the severity of pain increases, and as the score decreases, the severity decreases.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Aydın, Principal Investigator — esraaydin@gumushane.edu.tr-0456 2331149; Gülçin Avşar, Study Director — gulcin.avsar@atauni.edu.tr-0 442 2311584
Locations (2):
- Turkey (Türkiye) (2):
  - Ataturk University Faculty of Nursing, Erzurum, Centre
  - Gumushane Health Services Vocational School, Gümüşhane, Centre

IPD SHARING:
Plan to Share IPD: No